CLINICAL TRIAL: NCT03942458
Title: Pharmacokinetics and Pharmacodynamics of Vicagrel in Healthy Adult Subjects of Different CYP2C19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VCP1-Ⅰ-04
Record Dates: First submitted 2019-04-24; First posted 2019-05-08 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-03

CONDITIONS: Healthy Subjects; PK/PD
MeSH Terms: interventions — methyl 2-(2-acetoxy-6,7-dihydrothieno(3,2-c)pyridin-5(4H)-yl)-2-(2-chlorophenyl)acetate; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vicagrel (Experimental): Vicagrel 24mg loading followed by 6mg/day for 6 days
  Interventions: Drug: Vicagrel 6mg
- Clopidogrel (Active Comparator): Clopidogrel 300mg loading followed by 75mg/day for 6 days
  Interventions: Drug: Clopidogrel 75mg

INTERVENTIONS:
Drug: Vicagrel 6mg — Vicagrel 24mg loading followed by 6mg/day for 6 days
  Arms: Vicagrel
Drug: Clopidogrel 75mg — Clopidogrel 300mg loading followed by 75mg/day for 6 days
  Arms: Clopidogrel

SUMMARY:
This study is a single-center, randomized, open, two-cycle crossover, clopidogrel control, multiple dosing study. The aim was to evaluate the pharmacokinetic/pharmacodynamic behavior of different metabolites of CYP2C19 in healthy subjects. The study enrolled 48 patients, divided into three groups of CYP2C19 fast metabolite, middle metabolite, and slow metabolism, 16 cases in each group. All groups of subjects were administered for 7 days in the first cycle, once a day (loading dose on the first day, maintenance dose on other days), and entering the 14-day washout period after the end of the first cycle. The second cycle was entered, and the second cycle was administered for 7 days, once a day (the first day was given a loading dose, and the other days were given a maintenance dose). Blood was collected before and after administration of D1, D7, D22, and D28, and PK/PD was measured.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary signing of informed consent before the trial, and full understanding of the experimental content, process and possible adverse reactions;
* Subjects with ability and adherence to trial protocol;
* Subjects (including partners) voluntarily take effective contraceptive measures from screening to the last study drug administration within 6 months;
* Male and female aged 18-45,gender is unlimited (including 18 and 45 years old);
* Male Weight ≥50 kg, female Weight ≥ 45 kg, and BMI ranging from 18 to 28 kg/m2 (including critical values);
* Physical examination, normal or abnormal vital signs have no clinical significance (reference range of vital signs: systolic blood pressure 90-150 mmHg, diastolic blood pressure 50-95 mmHg, pulse 50-110 beats/min, body temperature 35.5-37.2 °C);
* CYP2C19 rapid metabolizers (CYP2C19*1/*1), or intermediate metabolizers (CYP2C19*1/*2, CYP2C19*1/*3), or poor metabolizers (CYP2C19*2/*2, CYP2C19*2/* 3, CYP2C19*3/*3).

Exclusion Criteria:

* More than 5 cigarettes per day 3 months before the trial;
* History of allergies or allergies to the drug (two or more drugs or food allergies);
* History of drug and/or alcohol abuse (14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine);
* Donate blood or massive blood loss (> 450 mL) within 3 months prior to formal screening;
* Take any drug that alters the activity of CYP450s within 28 days before the formal screening;
* Take any prescription, non-prescription, any vitamin or herbal medicine within 14 days of the formal screening;
* Take special diet (including dragon fruit, mango, grapefruit, etc.) within 2 weeks before the formal screening, or have strenuous exercise, or other factors affecting drug absorption, distribution, metabolism, excretion, etc.;
* Taking inhibitors or inducers of the CYP3A4, P-gp or Bcrp Currently, such as itraconazole, ketoconazole or dronedarone;
* Recently there have been major changes in diet or exercise habits;
* Taking other research drugs or participating in clinical trials within 3 months before taking the study drug;
* History of dysphagia or any gastrointestinal disease affecting drug absorption;
* Have any disease that increases the risk of bleeding, such as acute gastritis, stomach and duodenal ulcers, thrombocytopenic purpura, hemophilia, and so on;
* ECG abnormalities have clinical significance;
* Female subjects are in lactation or have a positive of pregnancy test;
* Clinical laboratory abnormalities have clinical significance or other clinically significant abnormalities (including but not limited to gastrointestinal, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental or cardiovascular and cerebrovascular diseases);
* Infectious diseases (two pairs of hepatitis B, hepatitis C antibodies, HIV, Treponema pallidum antibodies) have positive results;
* Acute disease or concomitant medication from the screening to the study;
* Taking chocolate, any food or drink with caffeine or jaundice-rich within 48 hours before taking the study drug;
* Any alcoholic product or alcohol breath test positive within 24 hours before taking the study drug;
* Urine drug test (morphine, marijuana) is positive;
* The investigator believes that there are other factors who are not suitable for participating in the test.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 1 day,7 days after taking drugs
  To evaluate the Peak Plasma Concentration (Cmax) after taking drugs
Area under the plasma concentration versus time curve (AUC) | 1 day,7 days after taking drugs
  To evaluate the AUC after taking drugsl
Time to maximum plasma concentration （Tmax） | 1 day,7 days after taking drugs
  To evaluate the Tmax after taking drugs
terminal half-life （T1/2） | 1 day,7 days after taking drugs
  To evaluate the T1/2 after taking drugs
inhibition of platelet aggregation | 1 day,7 days after taking drugs
  To evluate the inhibition of platelet aggregation assessed by Verifynow System after taking drugs

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China